CLINICAL TRIAL: NCT07290894
Title: Pembrolizumab Plus Lenvatinib in Vulvar Cancer Patients: MITO VULVA-01 Study.
Brief Title: Pembrolizumab Plus Lenvatinib in Vulvar Cancer Patients: MITO VULVA-01
Acronym: MITO VULVA-01
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MITO VULVA-01 2023-5091802400; 2023-509180-24-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-21; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Vulva Cancer
Keywords: vulvar cancer; pambrolizumab; lenvatinib; Phase II trial
MeSH Terms: conditions — Vulvar Neoplasms | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Intervention Model Description: pembrolizuma plus lenvatinib
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab+lenvatinib (Experimental): Pembrolizumab 200 mg + Lenvatinib 20 mg. Pembrolizumab will be administered up to 35 Cycles. Lenvatinib until disease progression or unaccetable toxicity
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib Capsules

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg IV infusion (30 minute) is administered at Day 1 of each 21-days cycle.Pembrolizumab will be administered up to 35 cycles.
Drug: Lenvatinib Capsules — .Lenvatinib 20 mg (two 10-mg capsules) QD will be taken orally with water (with or without food) in 21-day cycles at approximately the same time each day. On Day 1 of each Pembrolizumab cycle, Lenvatinib will be administered within 1 hour after Pembrolizumab.

SUMMARY:
MITO VULVA-1 is a prospective, single arm, multi-cohorts, phase II trial that aims to assess the activity and the safety of Lenvatinib plus Pembrolizumab in patients with vulvar cancer. 80 patients will be overall enrolled in the study.Three cohorts are planned

DETAILED DESCRIPTION:
In this study three cohorts are planned:

COHORT A: Locally advanced unresectable, treatments naïve, vulva carcinoma. Lenvatinib plus Pembrolizumab for 4 cycles. Then, in case of complete/partial clinical and/or pathological response Pembrolizumab monotherapy maintenance will be administered for a maximum of 35 cycles.

COHORT B: recurrent or de novo metastatic chemotherapy naïve, vulva carcinoma. These patients will receive Lenvatinib plus Pembrolizumab. Pembrolizumab will be administered for a maximum of 35 cycles and lenvatinb until PD, unacceptable toxicity, withdraw of consent.

COHORT C: recurrent or metastatic vulva carcinoma, in progression to a chemotherapy-based treatment or primary chemoradiation. These patients will receive Lenvatinib plus Pembrolizumab. Pembrolizumab will be administered for a maximum of 35 cycles, lenvatinb until PD, unacceptable toxicity, withdraw of consent.

Primary objectives To determine the activity (as assessed by objective response rate) and safety of Pembrolizumab plus Lenvatinib in vulvar cancer patients for each study cohorts.

Outcome Measures

* Objective response rate (ORR) defined as a complete response (CR) or partial response (PR) by the Investigator using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, in each single cohort (ORR will be evaluated after 4 cycles in Cohort A patients and on the whole treatment period in Cohort B and C patients)
* To evaluate the safety of 4 cycles of Pembrolizumab and Lenvatinib in vulvar cancer patients according to CTCAE (version 5.0) and PRO-CTCAE questionnaire in the overall study population (all the three cohorts together).

ELIGIBILITY:
Inclusion Criteria:

Target subject population Inclusion Criteria

1. Signed informed consent prior to any study specific procedure;
2. Female, age ≥ 18 years at time of signing informed consent;
3. Patients with histologically or cytologically confirmed unresectable squamous cell carcinoma, adenocarcinoma and mixed histology (adenosquamous) of the vulva, defined as:

   1. T2 or T3 primary tumors (N0-3, M0) not amenable to surgical resection by standard radical vulvectomy (Cohort A) OR
   2. recurrent or de novo metastatic chemotherapy-naive vulvar squamous cell carcinoma, adenocarcinoma and mixed histology (adenosquamous) of the vulva, (Cohort B) OR
   3. recurrent squamous cell carcinoma of the vulva after primary chemoradiation or patients with metastatic squamous cell carcinoma, adenocarcinoma and mixed histology (adenosquamous) of the vulva in progression to a chemotherapy-based treatment (Cohort C)
4. At least 1 measurable target lesion according to RECIST 1.1;
5. Patients must have a life expectancy ≥ 16 weeks;
6. ECOG performance status of 0 to 1;
7. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤140/90 mmHg at Screening and no change in antihypertensive medications within 1 week before the Cycle 1/Day 1;
8. Patient must provide formalin fixed paraffin embedded (FFPE), archival tumor samples, from primary tumor surgery or biopsy of primary tumor or metastases. The samples must be collected before any systemic treatment. (chemotherapy-naïve patients). A quality control analysis of samples will be performed before patient's enrollment. Only patients with adequate tumor samples will be enrolled.
9. Patient must be able to take oral medications;
10. Patients must have normal organ and bone marrow function measured as defined below:

    * Haemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5x ULN
    * Patients must have creatinine clearance estimated of ≥51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test: Estimated creatinine clearance = (140-age [years]) x weight (kg)(x F)a serum creatinine (mg/dL) x 72 (a where F=0.85 for females)
11. INR or PT aPTT/PTT ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants;
12. Patient is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

    1. Is not a Women of Childbearing Potential (WOCBP) or
    2. Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis), as described in Appendix 1 during the intervention period and for at least 4 months post pembrolizumab or 30 days post lenvatinib, whichever occurs last. The investigator should evaluate the potential for contraceptive method failure (ie, noncompliance, recently initiated) in relationship to the first dose of study intervention
13. A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before the first dose of study intervention; Note: If a urine test cannot be confirmed as negative (eg, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive;
14. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria

1. Patients with vulvar melanomas, sarcomas, vulvar Paget's disease, or basal cell carcinoma;
2. Patients diagnosed with early-stage vulvar cancer that, according to the Investigator, can be treated with upfront curative surgery;
3. Patients who have received any systemic anticancer therapy for vulvar cancer, anti-VEGF therapy, or any systemic investigational anticancer agent including radiotherapy (Cohort A and B); patients who have received any further systemic therapy for advanced disease after progression to a first-line platinum-based chemotherapy (Cohort C);
4. Received a live vaccine or live attenuated within 30 days of planned start of study treatment (Cycle 1/Day 1). Note: The killed virus vaccines (ie seasonal influenza vaccines for injection are allowed);
5. Has preexisting ≥Grade 3 gastrointestinal or non-gastrointestinal fistula;
6. Active infection (any infection requiring systemic treatment);
7. Subjects known to be positive for Human Immunodeficiency Virus (HIV);
8. Patients with known active hepatitis (i.e. Hepatitis B or C)

   * Active hepatitis B virus (HBV) is defined by a known positive HBV surface antigen (HBsAg) result. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible;
   * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA;
9. Subjects with a diagnosis of immunodeficiency or who are receiving systemic steroid therapy (dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medications;
10. Active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment;
11. Patients unable to swallow orally administered medication;
12. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment;
13. Major surgery within 3 weeks of starting study treatment and patients must have recovered from any effects of major surgery;
14. Breast feeding women;
15. Known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, (ie, without evidence of progression) for at least 4 weeks by repeat imaging (Note: The repeat imaging should be performed during study Screening.), clinically stable, and without requirement of steroid treatment for at least 14 days before the first dose of study intervention. Note: Participants with known untreated, asymptomatic brain metastases (ie, no neurological symptoms, no requirement for corticosteroids, no or minimal surrounding edema, and no lesion >1.5 cm) may participate but will require regular imaging of the brain as a site of disease;
16. Other malignancy unless curatively treated with no evidence of disease for ≥5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma
17. Prolongation of QTcF interval to ≥480 msec;
18. LVEF below of the institutional (or local laboratory), normal range, as determinated, by MUGA or ECHO;
19. Participation in another clinical study with an investigational product during the last 3 months;
20. Subjects who have not recovered adequately from any toxicity from other anti- cancer treatment regimens and/or complications from major surgery prior to starting therapy. Note: Withhold lenvatinib for at least 1 week prior to elective surgery. Do not administer for at least 2 weeks following major surgery and until adequate wound healing;
21. Significant cardiovascular impairment including: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction, cerebro vascular accident/stroke, within 12 months of the first dose of study drug, or cardiac arrhythmia associated with hemodynamic instability. Medically controlled arrhytmia would be permitted;
22. Bleeding or thrombotic disorders or subjects at risk for severe hemorrhage. Radiographic evidence of tumor invasion/infiltration of major blood vessels (e.g. carotid artery) or intratumoral cavitation. Note: The degree of major blood vessel should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy;
23. Radiographic evidence of tumor invasion/infiltration of major blood vessels (e.g. carotid artery) or intratumoral cavitation. Note: The degree of major blood vessel should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.
24. History of arterial tromboembolism within 12 months of start the study;
25. Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug;
26. Urine protein ≥1 g/24 hours. Note: Participants with proteinuria ≥2+ (≥100 mg/dL) on urine dipstick testing (urinalysis) will undergo 24-hour urine collection for quantitative assessment of proteinuria;
27. GI malabsorption or any other condition that might affect the absorption of Lenvatinib;
28. An allogenic tissue/solid organ transplant;
29. History of (noninfectious) pneumonitis/interstizial lung disease (ILD) that require steroids or current pneumonitis/ interstitial lung disease;
30. Known psychiatric disorder or substance abuse that would interfere with participant ability to cooperate with the requirement of the study.
31. Has received prior therapy with an anti-PD1, anti PD-L1 or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2031-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Objective Tumor Response Rate (ORR) | every 12 weeks from enrollment until disease progression (up to 72 months)
  Objective Tumor Response Rate (ORR) as defined by recist1.1 calculated as the proportion of patients achieving complete or partial response relative to total patients enrolled
Toxicity in the overall study population (all the three cohorts together). | At baseline during screening period (within 7 days prior to Cycle 1 Day 1), at day 1 of the first 4 cycles for patients in all cohorts. Cycle is defined as 21 days
  Toxicity rate is defined as the proportion of patients experiencing any grade AE accordingly to the NCI Common Terminology Criteria of Adverse Events (NCI CTC-AE) Version 5, relative to the total of patients receiving at least one cycle of treatment
  Toxicity will be evaluated also using Patient Reported Outcome Common Terminology Criteria of Adverse Events ( PRO-CTCAE) questionnaire.

SECONDARY OUTCOMES:
Progression free survival (PFS) | until progression of disease (up to 72 months)
  PFS is defined as the time elapsed from the date of randomization to the date of progression, as defined by investigators, or the date of death, whichever comes first. PFS will be evaluated in each single cohort
Overall Survival (OS) | up to 72 months
  OS is defined as the time elapsed from randomization to death due to any cause. OS will be evaluated in each single cohort. Patients alive at end of the study will censored at the date of the last follow-up contact
Toxicity | At the end of Cycle 5 day 1 ( each cycle is 21 days), until progression disease. (Up to 72 months)
  Description of overall safety of Pembrolizumab and Lenvatinib in patients who receive more than 4 cycles of treatment Toxicity rate is defined as the proportion of patients experiencing any grade AE accordingly to the NCI Common Terminology Criteria of Adverse Events (NCI CTC-AE) Version 5
  Toxicity will be evaluated also using Patient Reported Outcome Common Terminology Criteria of Adverse Events ( PRO-CTCAE) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, MD, PhD, Principal Investigator — National Cancer Institute,IRCCS, Fondazione G. Pascale, Naples , Italy
Locations (1):
- Nation Cancer Institute of Naples, Division of Medical Oncology - Uro-Gynecology Department, Naples, Napoli, Italy